CLINICAL TRIAL: NCT03289819
Title: A Phase II One-arm Open-label Neoadjuvant Study of Pembrolizumab in Combination With Nab-paclitaxel Followed by Pembrolizumab in Combination With Epirubicin and Cyclophosphamide in Patients With Triple Negative Breast Cancer
Brief Title: Neoadjuvant Pembrolizumab(Pbr)/Nab-Paclitaxel Followed by Pbr/Epirubicin/Cyclophosphamide in TNBC
Acronym: NIB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut fuer Frauengesundheit (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFG-NIB-01; 2016-003102-14 (EudraCT Number); U1111-1188-3915 (Other: WHO - (ICTRP))
Record Dates: First submitted 2016-10-11; First posted 2017-09-21 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Malignant Neoplasm of Breast
Keywords: TNBC; neoadjuvant chemotherapy; triple negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — pembrolizumab; 130-nm albumin-bound paclitaxel; Paclitaxel; Albumin-Bound Paclitaxel; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab/Nab-Paclitaxel (Experimental): This is a phase II, one-arm, open label neoadjuvant study of pembrolizumab in combination with nab-paclitaxel followed by pembrolizumab in combination with epirubicin and cyclophosphamide in patients with triple negative breast cancer.
  All patients will receive 12 cycles of weekly nab-paclitaxel intravenous (i.v.) 125 mg/m² body surface area (BSA) in combination with 4 cycles of pembrolizumab i.v. 200 mg q3w; followed by 4 cycles of epirubicin i.v. 90 mg/m² BSA and cyclophosphamide i.v. 600 mg/m² BSA, q3w in combination with 4 cycles of pembrolizumab i.v. 200 mg/kg q3w.
  After the 25th patient has started trial treatment, all further included patients will receive 1 additional cycle of pembrolizumab i.v. 200 mg q3w monotherapy before starting regular trial treatment.
  Clinical and bioptic tumor assessment will be performed after each treatment phase. Study treatment will be applied until state of the art surgery, onset of unacceptable toxicities, progression or withdrawal of consent.
  Interventions: Drug: Pembrolizumab; Drug: nab-paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Pembrolizumab — All patients will receive 12 cycles of weekly nab-paclitaxel intravenous (i.v.) 125 mg/m² body surface area (BSA) in combination with 4 cycles of pembrolizumab i.v. 200 mg q3w; followed by 4 cycles of epirubicin i.v. 90 mg/m² BSA and cyclophosphamide i.v. 600 mg/m² BSA, q3w in combination with 4 cycles of pembrolizumab i.v. 200 mg/kg q3w. After the 25th patient has started trial treatment, all further included patients will receive 1 cycle of pembrolizumab i.v. 200 mg q3w monotherapy followed by 12 cycles of weekly nab-paclitaxel intravenous (i.v.) 125 mg/m² body surface area (BSA) in combination with 4 cycles of pembrolizumab i.v. 200 mg q3w; followed by 4 cycles of epirubicin i.v. 90 mg/m² BSA and cyclophosphamide i.v. 600 mg/m² BSA, q3w in combination with 4 cycles of pembrolizumab i.v. 200 mg q3w.
  Other Names: Keytruda; MK-3475
Drug: nab-paclitaxel — All patients will receive 12 cycles of weekly nab-paclitaxel intravenous (i.v.) 125 mg/m² body surface area (BSA) in combination with 4 cycles of pembrolizumab i.v. 200 mg q3w; followed by 4 cycles of epirubicin i.v. 90 mg/m² BSA and cyclophosphamide i.v. 600 mg/m² BSA, q3w in combination with 4 cycles of pembrolizumab i.v. 200 mg/kg q3w.
  Other Names: nano-particle albumin bound (NAB) paclitaxel; Abraxane
Drug: Epirubicin — All patients will receive 12 cycles of weekly nab-paclitaxel intravenous (i.v.) 125 mg/m² body surface area (BSA) in combination with 4 cycles of pembrolizumab i.v. 200 mg q3w; followed by 4 cycles of epirubicin i.v. 90 mg/m² BSA and cyclophosphamide i.v. 600 mg/m² BSA, q3w in combination with 4 cycles of pembrolizumab i.v. 200 mg/kg q3w.
Drug: Cyclophosphamide — All patients will receive 12 cycles of weekly nab-paclitaxel intravenous (i.v.) 125 mg/m² body surface area (BSA) in combination with 4 cycles of pembrolizumab i.v. 200 mg q3w; followed by 4 cycles of epirubicin i.v. 90 mg/m² BSA and cyclophosphamide i.v. 600 mg/m² BSA, q3w in combination with 4 cycles of pembrolizumab i.v. 200 mg/kg q3w.

SUMMARY:
Despite its aggressiveness and high incidence, to date, no targeted therapies exist for the treatment of triple negative breast cancer (TNBC). Emerging evidence suggests a crucial role of tumor immunology on outcome for this entity. Checkpoint inhibitors like pembrolizumab, which target immune cells within the tumor, might therefore have an important impact on therapy response and outcome in these high risk patients. We propose a phase II study exploring pathological complete response and the safety of the combination of pembrolizumab and nab-paclitaxel as well as the combination of pembrolizumab with epirubicin and cyclophosphamide in the neoadjuvant setting for women with early TNBC. After completion of this study an extension will be determined.

DETAILED DESCRIPTION:
This is a multicenter, phase II, one-arm, open-label neoadjuvant study of pembrolizumab in combination with nab-paclitaxel followed by pembrolizumab in combination with epirubicin and cyclophosphamide (E/C) in patients with TNBC. Pathological complete response rate at the time of surgery is the primary objective of this study.

In approximately six large breast cancer centers in Germany 50 patients are planned to be enrolled. All patients will undergo state of the art staging and tumor assessments prior to study entry to assess eligibility for the present trial. Eligible and consented patients will receive 12 cycles of weekly nab-paclitaxel i.v. 125 mg/m² BSA q1w in combination with 4 cycles of pembrolizumab i.v. 200 mg q3w; followed by 4 cycles of epirubicin i.v. 90 mg/m² BSA and cyclophosphamide i.v. 600 mg/m² BSA, q3w in combination with 4 cycles pembrolizumab i.v. 200 mg q3w. After the 25th patient has started trial treatment, all further included patients will receive 1 cycle of pembrolizumab i.v. 200 mg q3w monotherapy followed by 12 cycles of weekly nab-paclitaxel intravenous (i.v.) 125 mg/m² body surface area (BSA) in combination with 4 cycles of pembrolizumab i.v. 200 mg q3w; followed by 4 cycles of epirubicin i.v. 90 mg/m² BSA and cyclophosphamide i.v. 600 mg/m² BSA, q3w in combination with 4 cycles of pembrolizumab i.v. 200 mg q3w. Clinical and bioptic tumor assessment will be performed after each treatment phase. Additional imaging, preferably with sonography, will be performed 6 weeks after initiation of taxane and anthracycline therapy to allow for early progress and response monitoring.

Study treatment will be applied until state of the art surgery, onset of unacceptable toxicities, progression or withdrawal of consent. A safety follow-up is planned 120 days after administration of the last dose of trial treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning of trial specific procedures.
2. Subject must be female and aged ≥ 18 years on day of signing informed consent.
3. ECOG(Eastern Cooperative Oncology Group) 0-1
4. Histologically confirmed, early TNBC determined by core biopsy of breast tumor lesion. ER and PR negativity are defined as ≤ 1% of cells expressing hormonal receptors via IHC (immuno-histochemistry) analysis. HER2(human epidermal growth factor receptor 2) negativity is defined as either of the following by local laboratory assessment: In situ hybridization (ISH) non-amplified (ratio ≤ 2.2), or IHC 0 or IHC 1+.
5. Measurable tumor lesion with a size of ≥ 1 cm assessed by sonography or magnetic resonance imaging (MRI) within ≤ 21 days prior to entry. In case of inflammatory disease the extent of inflammation will be measured.
6. Indication for chemotherapy.
7. Multicentric and/or multifocal disease, as well as synchronous bilateral breast cancer, is eligible as long as one measurable lesion meets all inclusion criteria. The investigator has to determine which lesion will be used for tumor evaluation before initiation of treatment.
8. Complete staging work up within 8 weeks prior to entry with no evidence of distant disease, including bilateral mammography, breast ultrasound, chest-X-ray (or chest CT-scan), liver ultrasound (or liver CT-scan or liver MRI) and bone scan.
9. Subjects must provide a core biopsy from tumor lesion at 3 time points (before, after first phase of treatment and at surgery) for central confirmation of TNBC status and biomarker analyses.
10. Adequate organ function, defined as:

    Absolute neutrophil count (ANC)≥ 1.5 x10³/μl, Hemoglobin ≥ 10.0 g/dl OR ≥ 6.2 mmol/l, Platelets ≥ 100 x10³/μl, Creatinine ≤ 1.5 x ULN OR GFR ≥ 30 ml/min, Total bilirubin ≤ 1.5 x ULN, AST (SGOT) and ALT (SGPT) ≤ 1.5 x ULN, Alkaline phosphatase ≤ 2.5 x ULN, International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN, Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN,
11. Female subjects of childbearing potential must have a negative urine pregnancy test within 72 hours prior to study entry and be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Concurrent participation in a study with an investigational agent/device or within 14 days of study entry.
2. Prior chemotherapy, radiation therapy or small molecule therapy for any reason.
3. Previous malignant disease being disease-free for less than 3 years (except in situ carcinoma of the cervix and basal cell carcinoma of the skin).
4. Pregnancy or lactation.
5. Prior therapy with an anti-PD1, anti-PD L1, anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g. CTLA-4, OX-40, CD137).
6. Active infection requiring systemic therapy.
7. History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
8. Active autoimmune disease or other diseases that requires systemic treatment with corticosteroids or immunosuppressive drugs (physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency is allowed).
9. History of primary or acquired immunodeficiency (including allogenic organ transplant).
10. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
11. Known history of following infections:

    1. Human immunodeficiency virus (HIV)
    2. History of acute or chronic Hepatitis B or Hepatitis C
    3. Has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted
12. Known congestive heart failure >NYHA I (New York Heart Association) and/or coronary heart disease, angina pectoris, previous history of myocardial infarction, uncontrolled or poorly controlled arterial hypertension (e.g. blood pressure >160/90 mmHg under treatment with two or more antihypertensive drugs), rhythm disorders with clinically significant valvular heart disease.
13. Preexisting motor or sensory neuropathy of a severity grade ≥ 2 by NCI CTCAE v4.0.
14. Known, pathogenic BRCA (breast cancer susceptibility gene) mutation. Note: testing is not mandatory for trial participation.
15. Any other condition in opinion of the investigator that would interfere with applied systemic treatment or other trial procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) rate | Pathological complete response will be assessed at final surgery for patients who received at least two cycles of Pembrolizumab. The rate will be assessed from 30 days until 120 days after last application of medication.
  Pathological complete response (pCR) rate, defined as the complete absence of all tumor cells (ypT0/ypN0), absence of invasive tumor (ypT0/is ypN0) and regression grades after study treatment. Pathological complete response is the primary endpoint of this trial and correlates especially well with disease-free survival and overall survival in patients with TNBC. Pathological complete response also serves as a surrogate marker for prognosis in TNBC

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | The adverse events will be assessed from first infusion until 120 days after last application of medication.
  The safety endpoints for the study will include rate of AE/SAEs and fatal SAEs, causality and outcome of AE/SAEs, rate of treatment discontinuations and reasons, changes in vital signs, laboratory values etc. Grading of AE/SAEs will be based on NCI CTCAE v4.0.
Clinical Response | Every 6 weeks from date of first medication administration until the date of first documented progression, surgery or date of death from any cause, whichever came first, assessed up to 120 days after last dose.
  To evaluate the efficacy of the treatment as measured by clinical response (objective response rate by 30 %) 6 weeks after the start of each sequential chemotherapy (nab-paclitaxel and E/C) and at the time of the surgery
EORTC QLQ-BR23 | Every two weeks from first administration of trial medication through study completion, up to 120 days after administration of last medication.
  To evaluate changes in health related quality of life (QoL) assessments from baseline in all subjects using the EORTC Breast Cancer-Specific Quality of Life Questionnaire (EORTC QLQ-BR23)
EORTC QLQ-C30 | Every two weeks from first administration of trial medication through study completion, up to 120 days after administration of last medication.
  To evaluate changes in health related quality of life (QoL) assessments from baseline in all subjects using Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)

OTHER OUTCOMES:
Tumor infiltrating lymphocytes (TILs) | Measured from biomaterial collected at baseline, 12 weeks after treatment initiation and at surgery.
  Tumor microenvironment prior to and during study treatment. TILs (stroma and intratumoral) in percent as assessed in Denkert et al. 2015, JCO.
Immunohistochemistry | Measured from biomaterial collected at baseline, 12 weeks after treatment initiation and at surgery.
  PD1 (Programmed cell death protein 1), PD-L1 (Programmed death-ligand 1), SPARC (Secreted protein acidic and rich in cysteine), Caveolin-1, TIM-3 (T-cell immunoglobulin mucin-3), Lag-3 (Lymphocyte-activation gene 3) will be assessed via immunohistochemistry in percentage of stained cells to total cell count and assesment of immunoreactive score (IRS) for each marker.
Tumor Immunogenicity | Measured from biomaterial collected at baseline, 12 weeks after treatment initiation and at surgery.
  Tumor immunogenicity characteristic measured via FACS of the following markers (CD45, CD3, CD4, CD8, CD14, CD19, CD25, CD56, CD127, CD197, HLA-DR, CD45RA, Ki67) in percent of positive cells to total cell count.
Mutational load | Measured from biomaterial collected at baseline, 12 weeks after treatment initiation and at surgery.
  Mutational load assessed by Next Generation Sequencing of Germline- and Tumor-DNA in mutations per megabases
Neoepitope Detection | Measured from biomaterial collected at baseline, 12 weeks after treatment initiation and at surgery.
  Amount of tumor neoepitopes assessed by Next Generation Sequencing comparing Germline- and Tumor-DNA. Neoepitopes are defined as mutations that lead to aminoacid changes and are found in tumor DNA only.
Cell-free RNA (cfRNA) | Measured from biomaterial collected at baseline, 12 weeks after treatment initiation and at surgery.
  Expression levels of specific tumor- and immune-related analytes in cfRNA will be measured by qPCR and possibly other methods and analyzed for correlations with subject outcomes.
Immune Status | Measured from biomaterial collected at baseline, 12 weeks after treatment initiation and at surgery.
  Peripheral Blood Mononuclear Cells will be collected from whole peripheral blood and sorted into subsets of T cells and myeloid cells by flow cytometry and then subjected to transcriptomic profilling by deep sequencing.
Circulation Metabolites | Measured from biomaterial collected at baseline, 12 weeks after treatment initiation and at surgery.
  Circulating metabolites of host and bacterial metabolites will be assessed in plasma using a multiplex 43-panel ELISA assay.
Microbial burden | Measured from biomaterial collected at baseline, 12 weeks after treatment initiation and at surgery.
  Viral, bacterial, fungal, helminth and parasite microbial burden will be assessed by Shotgun Deep Sequencing of cell-free RNA and DNA fragments in plasma.
Microbiome | Measured from biomaterial collected at baseline, 12 weeks after treatment initiation and at surgery.
  Stool microbiome will be assessed by Shotgun Deep Sequencing and analyzed for correlations with clinical outcome.
pCR rate after initiation boost | Pathological complete response will be assessed at final surgery for patients who received at least two cycles of Pembrolizumab. The rate will be assessed from 30 days until 120 days after last application of medication.
  To compare pCR rate in patients receiving a combination of pembrolizumab with nab-paclitaxel and epirubicin/cyclophosphamide chemotherapy and patients receiving 1 cycle of pembrolizumab monotherapy during an initiation boost followed by a combination of pembrolizumab with nab-paclitaxel and epirubicin/cyclophosphamide chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Fasching, MD, Prof., Study Chair — Department of Gynecology and Obstetrics, Erlangen University Hospital
Locations (4):
- Germany (4):
  - Department of Gynecology, Tübingen University Hospital, Tübingen, Baden-Wurttemberg
  - Department of Gynecology and Obstetrics, Erlangen University Hospital, Erlangen, Bavaria
  - Department for Gynecology and Obstetrics, Marienhospital Bottrop gGmbH, Bottrop, North Rhine-Westphalia
  - Department of Gynecology and Obstetrics, HELIOS Hospital Berlin Buch GmbH, Berlin

IPD SHARING:
Plan to Share IPD: No